CLINICAL TRIAL: NCT05588388
Title: IIT2022-05-Sankar-BELIEVE: Phase II Study of Bevacizumab in Combination With Chemoimmunotherapy and Maintenance Atezolizumab in Patients With Extensive Stage Small Cell Lung Cancer and Liver Metastases
Brief Title: Study of Bevacizumab in Combination With Chemoimmunotherapy and Atezolizumab in Patients With Extensive Stage Small Cell Lung Cancer and Liver Metastases
Acronym: BELIEVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kamya Sankar (Other)
Collaborators: Genentech, Inc. (Industry); University of Michigan (Other); VA Ann Arbor Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kamya Sankar, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022-05-Sankar-BELIEVE
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Extensive-stage Small-cell Lung Cancer; Liver Metastases
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): 1. Induction (ABCE): Atezolizumab 1200 mg, Bevacizumab 15 mg/kg, Carboplatin AUC5, Etoposide 100 mg/m2, given IV Q3weeks
  2. Maintenance (AB): Atezolizumab 1200 mg and Bevacizumab 15 mg/kg given IV Q3weeks for 1 year, or until disease progression, or unacceptable toxicity
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Addition of Bevacizumab to current standard of care treatment (atezolizumab, carboplatin and etoposide) followed by maintenance Bevacizumab plus Atezolizumab for patients with ES-SCLC with LM

SUMMARY:
This clinical trial aims to assess whether the addition of bevacizumab to atezolizumab and chemotherapy can improve response to treatment and progression-free survival in patients with extensive-stage small cell lung cancer (ES-SCLC) with liver metastases.

The main questions it aims to answer are:

* In patients with ES-SCLC with liver metastases, can bevacizumab in combination with atezolizumab and chemotherapy prolong the length of time that the cancer does not progress?
* Is bevacizumab safe and tolerable when combined with atezolizumab and chemotherapy in patients with ES-SCLC and liver metastases?

The study treatment includes two phases:

* Induction phase: bevacizumab will be administered in combination with atezolizumab and chemotherapy on a 21-day cycle for four cycles.
* Maintenance: atezolizumab and bevacizumab will be administered every 21 days for up to 12 months, or until unacceptable toxicity or disease progression.

Participants will undergo blood tests every 3 weeks and tumor assessments every 6 weeks.

DETAILED DESCRIPTION:
This is a phase II, open-label, multicenter, single-arm study designed to evaluate the efficacy and safety of bevacizumab plus atezolizumab plus carboplatin plus etoposide (ABCE) followed by bevacizumab plus atezolizumab (AB) maintenance in Extensive-Stage Small Cell Lung Cancer patients (ES-SCLC patients) with Liver Metastases (LM) who have received no prior systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability for subject to sign informed consent form and ability for subject to comply with the requirements of the study.
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group staging system), and radiographic confirmation of LM at diagnosis.
* Patients with history of EGFR mutant non-small cell lung cancer with histologically confirmed transformation to small cell lung cancer with presence of liver metastases, who are chemotherapy and immunotherapy naïve are eligible.
* No prior treatment for ES-SCLC. Note: patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of at least six months since the last chemotherapy, radiotherapy or chemoradiotherapy cycle prior to diagnosis of ES-SCLC
* Measurable disease per RECIST v1.1
* Asymptomatic patients with treated or untreated CNS lesions are eligible if there is no progression between completion of CNS-directed therapy and screening radiographic study, and the following criteria are met:

  * Metastases are limited to the cerebellum or supratentorial region (i.e., no metastases to the midbrain, pons, or medulla).
  * Presence of measurable disease outside the CNS per RECIST v1.1.
  * No history of intracranial hemorrhage or spinal cord hemorrhage.
  * No stereotactic radiotherapy or whole brain radiotherapy within 14 days prior to initiation of study treatment or neurosurgical resection within 28 days prior to initiation of study treatment.
  * Concurrent therapy of corticosteroids ≤ 10 mg of oral prednisone or equivalent and/or anticonvulsant therapy at stable dose.
* ECOG Performance Status of 0-2.
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 45 mL/min (calculated using the Cockcroft-Gault formula)
  * ANC ≥1.5 x 109/L (1500/µL) without granulocyte colony-stimulating factor support
  * Platelet count ≥ 100 x 109/L (100,000/µL) without transfusion
  * AST, ALT, and alkaline phosphatase (ALP) ≤ 5 x upper limit of normal (ULN), and serum bilirubin ≤ 1.5 x ULN
  * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN
  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* For patients who have positive hepatitis C antibody, HCV RNA must be performed at screening. For patients with a positive hepatitis C antibody with prior treatment or natural resolution who have negative HCV RNA are eligible. Patients with untreated hepatitis C may enroll if hepatitis is stable, and the patient is not at risk for hepatic decompensation. For those on concurrent HCV treatment, the HCV RNA level should be below the limit of quantification.
* Negative serum pregnancy test for women of childbearing potential.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, as defined below:

  * Women must remain abstinent or use an acceptable contraceptive method during the treatment period and for 5 months after the final dose of atezolizumab and 6 months after the final dose of bevacizumab.
  * A woman is considered to be of childbearing potential if she is post-menarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
  * Examples of acceptable contraceptive methods include, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during treatment with chemotherapy (i.e., carboplatin and etoposide) and for at least 6 months after the final dose of chemotherapy, atezolizumab and bevacizumab to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not adequate methods of preventing drug exposure.

Exclusion Criteria:

* History of leptomeningeal disease
* History of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to first dose of protocol therapy.
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)

  * Anti-hypertensive therapy to achieve these parameters is allowable.
* Evidence of tumor invading or abutting major blood vessels.
* Prior history of hypertensive crisis or encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* History of hemoptysis (≥one-half teaspoon of bright red blood per episode) within 1 month prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study enrollment) use of aspirin (> 325 mg/day) or treatment with dipyramidole, ticlodipine, clopidogrel, and clostazol
* Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for > 2 weeks prior to study enrollment

  * The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to enrollment.
  * Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR< 1.5 ×ULN and aPTT is within normal limits within 14 days prior to randomization. Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab
* History of abdominal or tracheosphageal fistula or gastrointestinal perforation within 6 months prior to study enrollment
* Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (refer to Appendix 12.5 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with rheumatoid arthritis who are on a stable pain regimen with symptom control.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:
* Rash must cover > 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of malignancy other than SCLC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate greater-than 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer treated surgically with curative intent.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

  o Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Known human immunodeficiency virus (HIV) infection. HIV-infected subjects on effective anti-retroviral therapy are eligible if the most recent viral load test performed within six months of screening (based on medical chart review) is negative.
* Known chronic hepatitis B
* Live, attenuated vaccines (e.g., FluMist®) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNFα agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after confirmation with the Principal Investigator has been obtained.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the bevacizumab formulation
* Currently taking or plan to take traditional herbal medicines.
* Treatment with investigational therapy within 28 days prior to initiation of study treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08-11 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
6- month Progression Free Survival (PFS) rate | Start of study treatment to 6-months
  Proportion of patients with first occurrence of disease progression or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From time of first dose until death or the first occurrence of disease progression whichever occurs first, assessed up to approximately 48 months
  Time from first dose of study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Overall Survival (OS) | From time of first dose until death from any cause, assessed up to approximately 48 months
  The length of time from date of first study treatment to death of any cause
Objective Response Rate | From time of first dose until time of best (maximal) response, assessed up to approximately 48 months
  Percent of patients who have either complete or partial response by CT/MRI imaging based on RECIST v1.1 criteria
Incidence of adverse events | From time of first dose until 90 days following the end of treatment, initiation of new systemic anti-cancer therapy, or death (whichever occurs first), assessed up to approximately 48 months
  Incidence of adverse events related to study treatment using CTCAE 5.0

OTHER OUTCOMES:
Tissue and blood based biomarkers | From baseline to approximately 15 months
  Identify tissue or blood based biomarkers that are associated with response to treatment with induction ABCE followed by maintenance AB in ES-SCLC patients with LM

CONTACTS AND LOCATIONS:
Overall Officials: Kamya Sankar, MD, Principal Investigator — Cedars-Sinai Cancer
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - V.A. Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No